CLINICAL TRIAL: NCT02785874
Title: Statin With Palliative Therapy for HCC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient for the fund
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N201603038
Record Dates: First submitted 2016-05-25; First posted 2016-05-30 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2016-05

CONDITIONS: HCC
MeSH Terms: interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Statin(Crestor) taken (Experimental): Subjects take Statin(Crestor) 10mg per day for a- year
  Interventions: Drug: Statin
- non Statin(Crestor) taken (No Intervention): non Statin(Crestor) taken as a reference for experimental group.

INTERVENTIONS:
Drug: Statin — Divide HCC patients into two groups under randomization, one is with Statin and the other is without Statin to verify whether Statin could prolong disease-free survival
  Arms: Statin(Crestor) taken

SUMMARY:
Statin is a preventive medicine for hepatitis B and hepatitis C which decreases the risk turning into liver cancer,however, the investigators also discovered that patients taking Statin live longer than patients who didn't take Statin in the incidence of liver cancer death cases.

DETAILED DESCRIPTION:
Most liver cancer patients did not accept the cure as the main objective of the treatment after diagnosis because they choose alternative therapies palliative based, such as hepatic arterial chemoembolization, chemotherapy and radiation therapy.

Statin is a preventive medicine for hepatitis B and hepatitis C which decreases the risk turning into liver cancer, yet the clinical effect for Statin is still unknown.

In a previous study of 20,220 liver cancer patients in health care database, the investigators discovered that patients taking Statin live longer than patients who didn't take Statin in the incidence of liver cancer death cases.

This study is a continuation of previous health insurance database studies for clinical trials to verify whether Statin could prolong disease-free survival role for palliative treatment of liver cancer.

ELIGIBILITY:
Inclusion Criteria:

1. >20 years old.
2. BCLC stage B , stage C and stage D

Exclusion Criteria:

1. Cancer diagnosis before HCC was conﬁrmed and incurable.
2. <20 years old, > 90years old.
3. Patients who are judged to be ineligible for study entry by the investigator or subinvestigator

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2016-10-01 (Actual); Study Completion 2016-11-01 (Actual)

PRIMARY OUTCOMES:
Overall Survival | Up to two year

CONTACTS AND LOCATIONS:
Overall Officials: Ming Shun Wu, Doctor, Study Chair — WanFangHospital
Locations (1):
- WanFangHospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No